CLINICAL TRIAL: NCT02743624
Title: Criteria Analysis for Ventilatory Support Adjustment of Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: tematicomusculoUTI
Record Dates: First submitted 2016-03-18; First posted 2016-04-19 (Estimated); Last update posted 2017-01-19 (Estimated); Status verified 2016-08

CONDITIONS: Acute Mechanical Ventilatory Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pressure Support Titration (Other): The analysis of the diagnostic accuracy of the breathing pattern variables, P 0.1 and the rate of tracheal muscle relaxation.
  Interventions: Procedure: Variation of the level of pressure support during the mechanical ventilation

INTERVENTIONS:
Procedure: Variation of the level of pressure support during the mechanical ventilation — The pressure support of the patient was changed form the baseline to 20 cmH20 and then stepwise decreased to 2 cmH20,

SUMMARY:
The indications for mechanical ventilation (MV) include excessive work of breathing, with or without evidence of respiratory muscle fatigue. The setting of the MV is still a challenge because it is based on criteria understudied, often subjective and observer-dependent. Despite several studies, to our knowledge has never been done before is the precise definition of the optimal range of ventilatory support. Novel and recognizable diagnostic techniques will be applied. No single parameter of the breathing pattern has good accuracy for the adjustment of ventilatory support. Non-invasive measures such as P0.1 and rate of muscle relaxation may have good accuracy for the adjustment of ventilatory support.

DETAILED DESCRIPTION:
Use of excessive pressure support

ELIGIBILITY:
Inclusion Criteria:

* patients under invasive mechanical ventilation for 48h
* patients without the objective of complete rest of the respiratory muscles. This decision will be on the discretion of the attending physician,
* spontaneous breathing,
* clinically stability.

Exclusion Criteria:

* Previous disease of the central nervous system that can lead to respiratory changes.
* Previous disease of the peripheral nervous system that can lead to respiratory changes
* Previous muscular disease.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2016-02; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Measuring muscular force | From the baseline ventilation to the minimum level of pressure support. Around 3 hours
  Muscular force measured by inspiratory force in centimeters of water (cmH2O)

SECONDARY OUTCOMES:
Measuring inspiratory drive | From the baseline ventilation to the minimum level of pressure support. Around 3 hours
  Inspiratory drive measured in cmH2O in the first 100 milliseconds of the inspiration
Measuring endurance | From the baseline ventilation to the minimum level of pressure support. Around 3 hours
  Endurance measured by the maximal relaxation rate (cmH2O/10ms)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Carvalho, Study Director — University of Sao Paulo
Locations (2):
- Brazil (2):
  - Hospital Clinicas Sao Paulo, São Paulo, São Paulo
  - Hearth Institute - University of Sao Paulo, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No